CLINICAL TRIAL: NCT06831084
Title: Acute Radiation Dermatitis After Adjuvant Radiotherapy for Breast Cancer Patients With the Use of Silver-Plated Technology: A Single Arm Phase II Trial
Brief Title: Acute Radiation Dermatitis After Adjuvant Radiotherapy for Breast Cancer Patients With the Use of Silver-Plated Technology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parul Barry (Other)
Collaborators: Bravida Medical (Unknown)
Responsible Party: Sponsor-Investigator, Parul Barry, Clinical Assistant Professor of Radiation Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCC 24-105
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Radiation Dermatitis Acute
Keywords: acute radiation dermatitis (ARD); Silver-plated technology (SPT) dressing; adjuvant radiotherapy (RT)
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Silver-Plated Technology dressing (Experimental): SPT dressing (Silverlon) worn for at least for 18 hours a day (removed while showering, bathing, and while having radiation therapy)
  Interventions: Device: Silver plated technology (SPT) dressing

INTERVENTIONS:
Device: Silver plated technology (SPT) dressing — Silver-plated technology (SPT) dressing technology is a wound dressing that has a permanently plated metallic surface, which provides the antimicrobial benefits of silver in the dressing without staining the skin and without increasing bioburden, reducing the development of acute radiation dermatitis (ARD).
  Other Names: Silverlon

SUMMARY:
Patients who are eligible to receive adjuvant whole breast radiotherapy with or without regional nodal irradiation as part of their care will be included in this study. Patients will use Silver-plated technology (SPT) dressing as directed per user instruction manual and change dressings weekly. Patients will continue to wear the SPT dressing for 2 weeks following completion of RT. The presence and severity of ARD will be recorded at the time of the weekly OTV and at one month after finishing the treatment.

DETAILED DESCRIPTION:
Adjuvant radiotherapy for breast cancer is standard in the setting of breast conserving therapy. The most common acute toxicity in those receiving breast radiotherapy is acute radiation dermatitis (ARD). This is not only disfiguring, but also painful and uncomfortable. No standard exists for the mitigation or treatment of ARD. Routinely, emollients and steroid based creams, including but not limited to, xeroform gauze, demeboro soaks, triple antibiotic cream, Silvadene, hydrocortisone, and mometasone creams are used. Steroid creams have been shown to change the skin microenvironment and also thin the skin - this is especially concerning as one of the primary goals of BCT is good to excellent cosmetic outcome. Mepitel dressings have been evaluated but are often cumbersome to use and difficult to apply accurately. Silver-plated technology (SPT) dressing, a novel skin dressing, has been shown to have anti-microbial effects thereby reducing the development of ARD. This prospective single arm phase II study will evaluate if SPT dressing reduces the incidence of grade 2 or higher ARD in breast cancer patients who are going to receive adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG ≤ 2
2. Male or female patients with breast cancer or breast carcinoma in situ who are recommended to receive adjuvant radiotherapy to the breast +/- regional lymph nodes or are planned to receive adjuvant radiotherapy to the chest wall and regional lymph nodes over 3 to 4 weeks.
3. Patients who will receive all of their RT at Magee Women's Hospital.
4. Agreeable to use of SPT dressing as directed (changing once weekly during RT and the additional 2 weeks following completion of RT).
5. Agreeable that any normal or physician recommended skin care regimen is to be used 1 hour prior to use of SPT dressing.
6. Agreeable to completion of assessments and skin checks and in person follow up at about 1 month following completion of RT.
7. Must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior RT to the breast +/- regional lymph nodes or prior RT to the chest wall and regional lymph nodes.
2. Contraindication to the application of SPT dressing (e.g. allergy).
3. Pregnancy/lactation or women of childbearing potential who are unable or unwilling to use adequate contraception during RT.
4. Planned RT course >4 weeks or <3 weeks.
5. Active connective tissue disorders/collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash in the area that will receive RT, systemic lupus erythematosis, or scleroderma.
6. Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent.
7. Known sensitivity or allergy to silver or nylon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or greater acute radiation dermatitis (ARD) | At 1 month post RT
  Proportion of patients grade 2 or higher acute radiation dermatitis (ARD). ARD is defined as skin changes ranging from faint erythema (reddening) and desquamation (peeling skin) to skin necrosis (death of skin cells) and ulceration, depending on the severity of the reaction that occur in those receiving breast cancer radiation therapy (RT) over 3-4 weeks.

SECONDARY OUTCOMES:
Use of advanced skin care products | Up to 1 month following completion of RT
  Proportion of patients receiving breast cancer radiation therapy (RT) over 3-4 weeks using advanced skin care products such as xeroform gauze, triple antibiotic cream, and/or Silvadene.
Patient satisfaction with silver-plated technology (SPT) dressing | At 1 month following completion of RT
  Proportion of patients receiving breast cancer radiation therapy (RT) over 3-4 weeks who are satisfied with SPT dressing as reported on the SPT Dressing Patient Satisfaction Survey. The SPT survey includes SPT individual attributes: Ease of prep and apply, Easy for patient use, Durable for repositioning, Patient Comfort, Wear time of 7 days, Patients overall satisfaction, Caregivers overall satisfaction, by "Satisfaction Levels (very satisfied, satisfied, neutral, dissatisfied, very dissatisfied) It also asks if the "Preferred Product" is the 'New' or 'Previous' product. There are four Yes/No questions also, inquiring as to whether the dressing provides relief when worn, able to be kept on before and after bathing, how many times cream was used to treat ARD, and understanding of directions for use. A scoring metric will be developed to quantify these results and analyze statistically. More 'satisfied' responses would indicate greater overall satisfaction with SPT.
Radiation Therapy (RT) Completion with use of silver-plated technology (SPT) | At 1 month following completion of RT
  Proportion of patients receiving breast cancer radiation therapy (RT) over 3-4 weeks using SPT dressing who complete RT in comparison to historical controls.
Silver-plated technology (SPT) Dressing ARD Visual Evaluation | At Baseline, At On Treatment Visits Weeks 1, 2, 3, 4, at 1 month
  The SPT Dressing ARD Visual Evaluation Form employs RTOG scoring: 0=No change over Baseline, 1=Follicular, faint or dull erythema, epilation, dry desquamation, decreased sweating, 2=Tender or bright erythema, patchy moist desquamation, moderate edema, 3=Confluent moist desquamation other than skin folds, pitting edema, 4=Ulceration, hemorrhage, necrosis. Total scores: 0-24, with higher scores indicating worse ARD.
Radiation-Induced Skin Reaction Assessment Scale (RISRAS) | At Baseline, At On Treatment Visits Weeks 1, 2, 3, 4, at 1 month
  The Radiation-Induced Skin Reaction Assessment Scale (RISRAS) and Distress Thermometer (DT) is a 31-point scale including 5 patient-reported domains (each scored 0-3) and 4 nurse-reported domains (each scored 0-4). The DT is solely patient-reported (0-10) and also queries specific factors contributing to distress. Patient questions include Tenderness, Discomfort, or Pain, Itch, Burning sensation, Skin reaction interfered with day to day activities, with 0-4 point ratings of "Not at all", "A little", "Quite a bit", "Very much". Nurse questions include presence/grading between 0-100% for Dry desquamation, Moist desquamation, Necrosis and coloring for Erythema between Normal and Deep Purple/Red (abnormal). Total scores: 0-36, with higher scores indicating worse ARD.

CONTACTS AND LOCATIONS:
Overall Officials: Parul N Barry, MD, Principal Investigator — UPMC Magee-Womens Hospital
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No